CLINICAL TRIAL: NCT05212467
Title: Amygdala and Insula Retraining (AIR) Program and HUS Internet Therapy Compared to Treatment as Usual in Bodily Stress Syndrome, Fibromyalgia, Post Covid-19, and Chronic Fatigue Syndrome (ME/CFS)
Brief Title: AIR-program and HUS Internet Therapy Compared to Treatment as Usual in Functional Disorders and Post Covid-19 Condition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Helena Liira, Chief Physician, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUS/2239/2021
Record Dates: First submitted 2022-01-24; First posted 2022-01-28 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Functional Disorders; Post Covid-19
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Patients are randomized to one of the three treatment groups
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AIR-program (Active Comparator): • The Amygdala and insula retraining program consists of novel brain retraining approaches focused on hypothetically interrupting and retraining the conditioned defensive hyper-stimulation of the sympathetic nervous system and aspects of the immune system by the amygdala and insula, to bring the brain and body back to homeostasis. It includes supportive techniques such as breathing, meditation, and neurolinguistic programming. The patients are invited to an online program of video session and eight weekly 2 h webinar sessions followed by three monthly sessions. The patients are assigned to do daily homework that takes approximately 15 to 20 min to complete
  Interventions: Behavioral: AIR-program; Behavioral: Treatment as usual
- HUS Internet therapy (Active Comparator): The HUS internet therapy for bodily stress syndromes (iHUSbss) includes psychoeducation about autonomic nervous system and of the effects of patient's own thinking and action on the nervous system. The exercises aim at relaxing the body, at novel ways to observe the symptoms, and at developing acceptance and self-compassion. The program includes exercises that are done regularly in everyday life.
  Interventions: Behavioral: HUS Internet therapy; Behavioral: Treatment as usual
- Treatment as usual (Placebo Comparator): The patients may have appointments with their physician, physiotherapist, or another health professional, and they may attend group interventions. If possible, medication is kept the same during the intervention and three months afterwards. If there is need to change the medication during the trial, the changes will be recorded. Appointments with health professionals and attendance in group interventions are monitored.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: AIR-program — This is a guided self management program that is added on the treatment as usual.
  Arms: AIR-program
Behavioral: HUS Internet therapy — This is a guided self management program that is added on the treatment as usual.
  Arms: HUS Internet therapy
Behavioral: Treatment as usual — The patients receive routine care from their physician which may include drugs, visits or rehabilitation

SUMMARY:
This study will compare an Amygdala and insula retraining (AIR) program to an internet therapy developed at Helsinki University Hospital. The study will be a multi-center randomized controlled trial. Study units will be recruited from the Network for Functional Disorders that is hosted by the HUS Clinic for Functional Disorders and potentially later from international collaborators. The trial will clarify whether internet-based non-drug based therapies are helpful in overcoming the central sensitization and the functional disabilities caused by these disorders.

DETAILED DESCRIPTION:
Functional disorders are a challenging group of conditions treated both in primary and secondary care. Recently, mounting evidence shows that central nervous system sensitization is one of the involved mechanisms, giving new treatment opportunities. There are self-management programs and internet therapies that aim at overcoming the central sensitization by creating new neural networks in the brain. This study aims to test whether an Amygdala and insula retraining (AIR) program compared to an internet therapy developed at HUS (Helsinki University Hospital) and treatment as usual (TAU) is effective in the treatment of functional disorders, fibromyalgia, long Covid, and chronic fatigue syndrome (ME/CFS).

The investigators will perform a multi-center randomized controlled trial in volunteering health units and with volunteering patients aiming at 360 patients altogether. The physicians in charge of the patients will be recruited from the Network for Functional Disorders launched by the novel clinic at HUS. The participating centers will receive an introduction in functional disorders, the underlying mechanisms, and treatment opportunities.

For functional disorders, this study applies the ICD-11 primary care code of Bodily stress syndromes (BSS), which covers fibromyalgia, irritable bowel syndrome, multiple chemical sensitivities, and other, both single system and multiorgan functional disorders. In addition, for patients with fibromyalgia, chronic fatigue symptoms, and Post Covid-19 condition, we will apply specific diagnostic criteria. Both primary and secondary care treatment units that manage these disorders can recruit patients.

The studied interventions are an Amygdala and insula retraining (AIR) program and an internet therapy developed at HUS, and patients receive usual care in addition to these interventions. The third study arm consists of treatment as usual for six months after which the patients receive the AIR program or the internet therapy if they so wish. When the participating physicians consider that a patient could benefit from a self-management program, they introduce the trial to the patient. The consenting patient fills in a baseline survey and is followed up at 3, 6, and 12 months with the help of the HUSeCRF (online surveys at the HUS electronic Case Report Form), or research nurse's interviews.

This study will give new insight into the opportunities of self-management programs in the treatment of bodily stress syndromes, fibromyalgia, Post Covid-19, and ME/CFS. The investigators will find out whether the training programs increase patients' functional ability and quality of life as measured on a scale from 0 to 10. These scales and functional ability as measured by WHODAS 2.0 serve as main outcome measures for this study. This trial is the first large-scale randomized trial that assesses these methods developed to overcome the central sensitization of brain. The results will have an impact on the management of these common and often debilitating conditions.

ELIGIBILITY:
Inclusion Criteria:

* • The criteria of bodily stress syndrome, fibromyalgia, chronic fatigue syndrome, or long Covid fulfilled AND

  * Diagnostic examinations have ruled out the potential somatic reasons for the symptoms AND
  * Disabling symptoms have lasted at least 3 months AND
  * Patient is willing to receive a psychoeducation or brain retraining intervention.

Exclusion Criteria:

* • Patients for whom participation could be overly demanding because of physical constraints (for example, patients who cannot write because of dystonia or bedridden patients)

  * Patients with presence of severe psychiatric and severe somatic disorders, e.g. moderate or severe depression or newly onset cancer for which the study could be overly strenuous.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2022-01-31 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in functional ability as measured by the WHODAS2.0 instrument at six months. | 3, 6 and 12 months

SECONDARY OUTCOMES:
Change from baseline in quality of life as measured by EUROHIS-8 | 3, 6 and 12 months
Change from baseline in health related quality of life as measured by 15D | 3, 6 and 12 months
Change from baseline in symptoms as measured by SSD-12 and PHQ-15 | 3, 6 and 12 months
Change from baseline in depression as measured by PHQ-9 | 3, 6 and 12 months
Change from baseline in anxiety as measured by GAD-7 | 3, 6 and 12 months
Change in sleep as measured by ISI | 3, 6 and 12 months
Change in resilience as measured by Resilience Scale-14 | 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- Finland (2):
  - Clinic for Functional Disorders, HUS, Helsinki
  - Clinic for Long Covid, HUS, Helsinki

IPD SHARING:
Plan to Share IPD: Undecided
We have applied for EU Horizon funding and may share data in that project.

REFERENCES:
- [Derived] Vangelova-Korpinen V, Liira H, Kurki SN, Sainio M, Malmivaara A, Kanerva M, Stenberg JH, Varonen M, Venalainen M, Vuorela P, Arokoski J. Effectiveness of mindfulness-based online therapy or internet-delivered cognitive behavioral therapy compared with treatment as usual among patients with persistent somatic symptoms: Protocol for a randomized controlled trial. PLoS One. 2025 Feb 12;20(2):e0316169. doi: 10.1371/journal.pone.0316169. eCollection 2025. PMID 39937805